CLINICAL TRIAL: NCT02308722
Title: A Phase I Trial of Pre-operative, Margin Intensive, Stereotactic Body Radiation Therapy for Pancreatic Cancer
Brief Title: SBRT Pre-operatively for Pancreatic Cancer
Acronym: SPARC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oncology Clinical Trials Office (Unknown); Centre for Statistics in Medicine (Other); CRUK/MRC Oxford Institute for Radiation Oncology (Unknown); University of Leeds (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_054; 18496 (Other: UKCRN ID); 14138956 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2021-10-07 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Neoplasms
Keywords: Borderline resectable
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5-fraction stereotactic body radiation therapy (Experimental): See intervention
  Interventions: Radiation: 5-fraction stereotactic body radiation therapy

INTERVENTIONS:
Radiation: 5-fraction stereotactic body radiation therapy — The investigators expect to need a maximum of 3 dose levels investigating dose to the area at risk of involved resection lines and to the tumour bed to assess the tolerability of SBRT in this setting.
  Patient entry will commence at level 1. There is the option to de-escalate to Level -1 should 2 or more DLTs be observed at the starting level. SBRT will not be escalated above level 3.
  Level -1:
  Tumour (PTV) 6Gy/# (total dose 30Gy). Area at risk of R1 (PTV_R) 8Gy/# (total dose 40Gy)
  Level 1:
  Tumour (PTV) 6Gy/# (total dose 30Gy). Area at risk of R1 (PTV_R) 9Gy/# (total dose 45Gy)
  Level 2:
  Tumour (PTV) 6.5Gy/# (total dose 32.5Gy). Area at risk of R1 (PTV_R) 9.5Gy/# (total dose 47.5Gy)
  Level 3:
  Tumour (PTV) 7Gy/# (total dose 35Gy). Area at risk of R1 (PTV_R) 10Gy/# (total dose 50Gy)

SUMMARY:
In this study the investigators are testing if the addition of Stereotactic Body Radiation therapy (SBRT) prior to surgery improves surgical outcome in patients with borderline resectable or resectable pancreatic cancer (BRPC).

DETAILED DESCRIPTION:
This is a single arm prospective phase I dose escalation radiation study investigating 5-fraction stereotactic radiotherapy prior to planned surgical resection in borderline resectable or resectable pancreatic cancer.

Surgical resection is the only potentially curative technique for managing pancreatic cancer. However more than 80% of patients present with disease that cannot be cured with surgical resection. Negative margin (R0 resection), tumour size, absence of lymph nodes metastases are the strongest prognostic indicators for long term survival.

Stereotactic body radiation therapy (SBRT) is a radiation technique for pancreatic cancer where an ablative dose of radiotherapy (RT) can be delivered to a small volume targeting the at risk surgical margin in a short time (1 week versus 5-6 weeks for standard radiotherapy), achieving much higher biologically equivalent dose (BED) (100Gy versus 50Gy) than conventionally fractionated radical RT. The short time of delivery and minimal acute toxicity makes this an attractive treatment option in BPRC as offers the opportunity to integrate systemic treatment. With standard fractionation schedules larger volumes of normal tissue are usually irradiated than with SBRT and an effective dose is limited by toxicity despite the use of Intensity Modulated RT.

This study builds on the current evidence base in SBRT pancreas, which has so far been largely used in the locally advanced setting with promising results and aims to take it a step further. This study aims to test the safety and benefit of pre-operative SBRT, delivering very high local doses to the at risk surgical margin which is usually around the main vessels in the retroperitoneum. The concept of margin-intensive therapy is novel, and aims to deliver a higher radiation dose while limiting toxicity to organs at risk.

ELIGIBILITY:
Inclusion Criteria:

1. Borderline resectable localised tumour of the pancreatic head/uncinate process/body as per NCCN Guidelines (tumours of the tail of pancreas are not eligible for inclusion) or operable tumour in contact with vein (SMV or PV) not causing distortion or narrowing as defined by CT +/- MRI +/- PET criteria within 28+/- 7 days prior to trial entry de novo or following chemotherapy.
2. Histologically proven pancreatic ductal adenocarcinoma or cytological proven pancreatic malignancy.
3. Able to undergo biliary drainage using a stent.
4. Deemed fit and suitable for surgical resection.
5. No overt metastases or uncertain status with investigations suspicious of possible metastatic disease (e.g. small equivocal pulmonary nodule(s)).
6. Male or female, Age >= 16 years.
7. Life expectancy of at least 6 months.
8. ECOG performance status 0- 1
9. The patient is willing and able to comply with the protocol for the duration of the study, and scheduled follow-up visits and examinations.
10. Written (signed and dated) informed consent and be capable of co-operating with protocol.
11. Haematological and biochemical indices within defined ranges.

Exclusion Criteria:

1. Distant metastatic disease or local disease that cannot be encompassed in the SBRT field.
2. History of previous or concurrent malignancy diagnoses for which the expected prognosis is likely to be worse than that for the current diagnosis of pancreatic cancer (excludes for example: e.g. localised prostate cancer, early colorectal cancer, early breast cancer, curatively-treated basal cell carcinoma of skin, carcinoma in situ of cervix; curatively treated cancer of other sites who are recurrence free for >3 years).
3. Serious medical or psychological condition precluding trial intervention.
4. Previous upper abdominal or right chest wall radiotherapy where 30% of the liver has received >15Gy.
5. PPregnancy. Pregnant or breast-feeding women are ineligible. Women of childbearing potential must use effective methods of contraception.
6. Any other psychological, social or medical condition, physical examination finding or laboratory abnormality that the Investigator considers makes the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of the trial results.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 30 days from SBRT day 1
  The maximum tolerated dose (MTD) is defined as the highest dose of margin-intensive SBRT delivered pre-operatively at which no more than 1 of 6 patients or 0 of 3 patients experiences a dose limiting toxicity (DLT)

SECONDARY OUTCOMES:
Definitive resection rate | Surgery
R0/R1/R2 resection margin rates | Pathological specimen evaluated at surgery
Rate of pathological complete response | Pathological specimen evaluation post operation
Any Late GI AE/other AE > grade 2 CTCAE v4.03 | >1 month to 6 months post-surgery
Overall survival and progression free survival at 12 and 24 months post D1 SBRT | 12 and 24m FU

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Maria A Hawkins, MD FRCR MRCP, Principal Investigator — University of Oxford
Locations (5):
- United Kingdom (5):
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - St James' Hospital, Leeds
  - Northern Centre for Cancer Care, The Freeman Hospital, Newcastle
  - City Hospital, Nottingham
  - The Churchill Hospital, Oxford University Hospitals Trust, Oxford

REFERENCES:
- [Result] Holyoake DLP, Robinson M, Silva M, Grose D, McIntosh D, Sebag-Montefiore D, Radhakrishna G, Mukherjee S, Hawkins MA. SPARC, a phase-I trial of pre-operative, margin intensified, stereotactic body radiation therapy for pancreatic cancer. Radiother Oncol. 2021 Feb;155:278-284. doi: 10.1016/j.radonc.2020.11.007. Epub 2020 Nov 18. PMID 33217498
- [Derived] Holyoake DL, Robinson M, Grose D, McIntosh D, Sebag-Montefiore D, Radhakrishna G, Patel N, Partridge M, Mukherjee S, Hawkins MA. Conformity analysis to demonstrate reproducibility of target volumes for Margin-Intense Stereotactic Radiotherapy for borderline-resectable pancreatic cancer. Radiother Oncol. 2016 Oct;121(1):86-91. doi: 10.1016/j.radonc.2016.08.001. Epub 2016 Aug 9. PMID 27519585
- See also: Results paper — https://pubmed.ncbi.nlm.nih.gov/33217498/